CLINICAL TRIAL: NCT05105347
Title: Efficacy and Safety of Adalimumab Plus Medium Dose Oral Glucocorticosteroid for Refractory Behçet's Uveitis, Compared With Adalimumab Plus High Dose Oral Glucocorticosteroid, a Non-inferior, Multi-center, Randomized Controlled Trial.
Brief Title: Efficacy and Safety of Adalimumab Plus Medium Dose Oral Glucocorticosteroid for Refractory Behçet's Uveitis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 42-ZS-2925
Record Dates: First submitted 2021-10-19; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis | interventions — Adalimumab; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medium dose group (Adalimumab plus medium dose oral glucocorticosteroid) (Experimental): Patients will be given adalimumab with 30mg daily prednisone or equivalent with a fixed slow tapering plan.
  Interventions: Drug: Adalimumab plus different doses of oral glucocorticosteroid
- High dose group (Adalimumab plus high dose oral glucocorticosteroid) (Active Comparator): Patients will be given adalimumab with 60mg daily prednisone or equivalent with a fixed slow tapering plan.
  Interventions: Drug: Adalimumab plus different doses of oral glucocorticosteroid

INTERVENTIONS:
Drug: Adalimumab plus different doses of oral glucocorticosteroid — A loading dose of 80mg adalimumab will be given subcutaneously and then change to 40mg adalimumab every two weeks. Medium dose oral glucocorticosteroid (30mg/d prednisone or equivalent) will be given to the experimental dose group and high dose oral glucocorticosteroid (60mg/d prednisone or equivalent) will be given to the high dose group.
  Other Names: Humira, prednisone

SUMMARY:
This study is a multi-center randomized non-inferiority study that aims to observe the short-term (3 months) efficacy and safety of adalimumab plus medium-dose glucocorticosteroid (30mg/d prednisone or equivalent) with slow tapering for recurrent Behçet's uveitis (BU) attack compared with adalimumab plus high-dose glucocorticosteroid (60mg/d prednisone or equivalent) with slow tapering.

DETAILED DESCRIPTION:
According to the most recent European League Against Rheumatism (EULAR) recommendation, patients presenting with an initial or recurrent episode of acute sight-threatening uveitis should be treated with high-dose glucocorticoids, infliximab or interferon-α. Adalimumab, another TNFα antagonist, is also considered as an alternative for infliximab and have proved its efficacy in several RCTs in the treatment of non-infectious intermediate, posterior and pan-uveitis. As higher dose glucocorticosteroid have greater side effects, this study aims to evaluate the non-inferior efficacy and safety of adalimumab plus medium-dose glucocorticosteroid compared with adalimumab plus high-dose glucocorticosteroid (and slow tapering) for recurrent posterior or pan-uveitis attack of Behcet's uveitis. Refractory BU is defined as relapse of posterior or panuveitis with at least 10mg daily prednisone (or equivalent). The acute attack will be controlled with adalimumab (80mg once, 40mg q2w thereafter) plus medium dose initial oral glucocorticosteroid (30mg daily prednisone or equivalent) in the "medium dose" group or plus high dose oral glucocorticosteroid (60mg daily prednisone or equivalent) in the "high dose" group with fixed tapering protocols. Patients will be followed up at 2w, 4w, 8w, and 12w after initiation of treatment. The primary endpoint is the inflammatory control rate. Secondary endpoints are BCVA, vascular leakage score on fundus fluorescein angiography (FFA), BOS 24 score and uveitis deterioration rate. The safety profiles of both groups will be also monitored.

ELIGIBILITY:
Inclusion Criteria:

* Behçet's disease (BD) patients fulfilling the International Criteria for Behçet's disease (ICBD) published in 2013 with recent recurrence of pan- or posterior uveitis
* The patient should be on ≥10mg/d oral prednisone or equivalent

Exclusion Criteria:

* Previous treatment with TNFα inhibitors within 3 months
* Pregnancy, breast feeding women
* Malignancy
* Heart failure
* Demyelinating diseases
* Renal impairment (creatinine > 1.5 mg/dl)
* Depression or other psychic disorders
* History of acute or chronic inflammatory joint or autoimmune disease
* Patients with severe extra-ocular involvement other than oral/genital ulcer and skin involvement
* Organ or bone marrow transplant recipient, cardiac failure > NYHA III
* Acute liver disease with ALT or SGPT 2x above normal
* White blood cell count < 3500/mm^3
* Platelet count < 100000/mm^3
* Hgb < 8.5g/dl
* T-SPOT TB: ≥200 SFCs per 10^6 PBMC
* Active peptic ulcer, systemic or local infection, moderate to severe osteoporosis or other contraindications of intermediate dose corticosteroids
* Other severe ocular diseases or intraocular surgery within 3 months
* Media opacity precluding a clear view of the fundus
* Positive screen test for HBV, HCV, HIV infection or syphilis
* Body weight <45 kg
* Alcohol abuse or drug abuse
* Mental impairment
* Uncooperative attitude

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-11-10 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Uveitis control | 3 months
  Inflammation control according to SUN criteria (two steps decrease of anterior chamber cell or vitreous haze or decreased to zero) or active retinal lesion recession with vitreous haze less than 0.5 grade

SECONDARY OUTCOMES:
Best corrected visual acuity (BCVA) | 3 months
  BCVA was transformed into logMar form
Extent of vascular leakage | 3 months
  Vascular leakage was quantified based on the method developed by the Angiography Scoring for Uveitis Working Group (ASUWOG), in which vascular leakage in the posterior pole and in each peripheral quadrant was scored 1 if limited
BOS 24 score | 3 months
  BOS 24 scoring system refers to article "Behc et's disease ocular attack score 24: evaluation of ocular disease activity before and after initiation of infliximab
Uveitis deterioration | 3 months
  Inflammation deterioration according to SUN criteria (two steps increase of anterior chamber cell or vitreous haze or increases to grade 4) or new active retinal lesions or new onset of retinal vasculitis

IPD SHARING:
Plan to Share IPD: Undecided
email contact person if needed

REFERENCES:
- [Background] Jaffe GJ, Dick AD, Brezin AP, Nguyen QD, Thorne JE, Kestelyn P, Barisani-Asenbauer T, Franco P, Heiligenhaus A, Scales D, Chu DS, Camez A, Kwatra NV, Song AP, Kron M, Tari S, Suhler EB. Adalimumab in Patients with Active Noninfectious Uveitis. N Engl J Med. 2016 Sep 8;375(10):932-43. doi: 10.1056/NEJMoa1509852. PMID 27602665
- [Background] Levy-Clarke G, Jabs DA, Read RW, Rosenbaum JT, Vitale A, Van Gelder RN. Expert panel recommendations for the use of anti-tumor necrosis factor biologic agents in patients with ocular inflammatory disorders. Ophthalmology. 2014 Mar;121(3):785-96.e3. doi: 10.1016/j.ophtha.2013.09.048. Epub 2013 Dec 17. PMID 24359625
- [Background] Vallet H, Riviere S, Sanna A, Deroux A, Moulis G, Addimanda O, Salvarani C, Lambert M, Bielefeld P, Seve P, Sibilia J, Pasquali J, Fraison J, Marie I, Perard L, Bouillet L, Cohen F, Sene D, Schoindre Y, Lidove O, Le Hoang P, Hachulla E, Fain O, Mariette X, Papo T, Wechsler B, Bodaghi B, Rigon MR, Cacoub P, Saadoun D; French Behcet Network. Efficacy of anti-TNF alpha in severe and/or refractory Behcet's disease: Multicenter study of 124 patients. J Autoimmun. 2015 Aug;62:67-74. doi: 10.1016/j.jaut.2015.06.005. Epub 2015 Jul 8. PMID 26162757
- [Background] Kaburaki T, Namba K, Sonoda KH, Kezuka T, Keino H, Fukuhara T, Kamoi K, Nakai K, Mizuki N, Ohguro N; Ocular Behcet Disease Research Group of Japan. Behcet's disease ocular attack score 24: evaluation of ocular disease activity before and after initiation of infliximab. Jpn J Ophthalmol. 2014 Mar;58(2):120-30. doi: 10.1007/s10384-013-0294-0. Epub 2014 Jan 31. PMID 24482146